CLINICAL TRIAL: NCT05968001
Title: Efficacy and Safety of Obinutuzumab in Chinese Patients With Indolent Non-Hodgkin's B-cell Lymphoma in the Real-World.
Brief Title: Obinutuzumab in Chinese Real-world Patients With iNHL
Status: Not yet recruiting | Type: Observational
Sponsor: Affiliated Hospital of Nantong University (Other)
Responsible Party: Principal Investigator, Wenyu Shi, Director, Department of Oncology, Affiliated Hospital of Nantong University
Other Study IDs: JCLG-23-04
Record Dates: First submitted 2023-07-23; First posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Lymphomas Non-Hodgkin's B-Cell
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — obinutuzumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cohort 1: the younger cohort (aged ≥ 18 and < 60 years at the start of treatment)
  Interventions: Drug: Obinutuzumab
- Cohort 2: the older cohort (aged ≥ 60 years at the start of treatment)
  Interventions: Drug: Obinutuzumab

INTERVENTIONS:
Drug: Obinutuzumab — obinutuzumab (G)-contained regimens, including GB, G-CHOP, and G-CVP.

SUMMARY:
This study aims to assess the clinical efficacy and safety of obinutuzumab in Chinese patients with indolent non-Hodgkin B-cell Lymphoma (predominantly Follicular lymphoma and Marginal zone lymphoma) in a real-world setting.

DETAILED DESCRIPTION:
This study was a prospective, multicenter, non-interventional, real-world study. The study will be divided into two cohorts: Cohort 1 is the younger cohort (aged ≥ 18 and < 60 years at the start of treatment); Cohort 2 is the older cohort (aged ≥ 60 years at the start of treatment). Patients in this study will receive obinutuzumab-contained regimens according to the investigators' clinical opinion.

ELIGIBILITY:
Inclusion Criteria:

* Age: Age ≥ 18 years at the start of treatment;
* Be diagnosed with grade 1-3a follicular Lymphoma, Marginal zone lymphoma;
* Previously untreated or relapsed or refractory patients;
* Patients who started treatment with otuzumab between June 2021 and April 2023.

Exclusion Criteria:

* Patients currently participating or planning to participate in any interventional clinical trial;
* Patients who, in the opinion of the investigator, are Discomfort for any other reason to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with FL and MZL who started treatment with otuzumab between June 2021 and April 2023.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-07-20 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2026-07-20 (Estimated)

PRIMARY OUTCOMES:
Efficacy Endpoints | 12 months
  The best objective response rate (ORR), and CR rate; ORR and CR rate at the end of treatment; DCR, DoR, TTNT, PFS, DFS, and OS.

SECONDARY OUTCOMES:
Safety Endpoints | 12 months
  All AEs, SAEs, Grade 3 AEs, and all other safety variables, including vital signs, Physical examination results, and laboratory parameters.

OTHER OUTCOMES:
Exploratory Endpoints | 12 months
  Subgroup analyses will be performed for some special populations, such as in high-risk patients

CONTACTS AND LOCATIONS:
Locations (25):
- China (25):
  - Changzhou No.2 People's Hospital, Changzhou, Jiangsu
  - The First People's hospital of Changzhou, Changzhou, Jiangsu
  - Huai'an First People's hospital, Huai'an, Jiangsu
  - Jiangyin People's Hospital, Jiangyin, Jiangsu
  - Jingjiang People's Hospital, Jingjiang, Jiangsu
  - The first people's hospital of Lianyungang, Lianyungang, Jiangsu
  - The second people's hospital of Lianyungang, Lianyungang, Jiangsu
  - Jiangsu Province Hospital of Chinese Medicine, Nanjing, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Nanjing Jiangning Hospital, Nanjing, Jiangsu
  - Nantong Tumor Hospital, Nantong, Jiangsu
  - Affiliated Hospital of Nantong University, Nanyang, Jiangsu
  - The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Jiangsu Taizhou People's Hospital, Taizhou, Jiangsu
  - Affiliated Hospital of Jiangnan University, Wuxi, Jiangsu
  - Wuxi People's Hospital, Wuxi, Jiangsu
  - Wuxi Second People's Hospital, Wuxi, Jiangsu
  - Yancheng No.1 People's Hospital, Yancheng, Jiangsu
  - Yancheng Third People's Hospital, Yancheng, Jiangsu
  - Subei People's Hospital, Yangzhou, Jiangsu
  - Yixing People's Hospital, Yixing, Jiangsu
  - Zhangjiagang First People's Hospital, Zhangjiagang, Jiangsu
  - Affiliated Hospital of Jiangsu University, Zhenjiang, Jiangsu
  - Zhenjiang First People's Hospital, Zhenjiang, Jiangsu

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, ICF, CSR
Time Frame: starting 6 months after publication
Access Criteria: IPD could be shared by contacting the corresponding author via email after publication.